CLINICAL TRIAL: NCT03687580
Title: Effectiveness and Safety of a Home-Use Low Level Laser Therapy Device As an Adjunct to Standard Treatment Compared to Standard Treatment Alone, for Diabetic Foot Ulcers: a Double Blind, Randomized, Sham-Controlled Clinical Study
Brief Title: Laser Therapy for At-Home Treatment of Diabetic Foot Ulcers - Canada
Acronym: LLL&DIAB-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scarborough Rouge Hospital (Other)
Responsible Party: Principal Investigator, Rose Raizman, Principle Investigator, Scarborough Rouge Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUR-18-010
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Photobiomodulation; Low-Level Laser Therapy; over the counter
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single center, Prospective, Double Blind, Randomized, Sham-Controlled, Parallel Group, Superiority comparison
Who Masked: Participant, Care Provider, Investigator
Masking Description: The active and sham devices are externally identical and emit the same guiding light. The only difference is that the sham does not emit the therapeutic near infrared rays. However, since near infrared laser light is invisible to the human eye, the treatment allocation cannot be determined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- B-Cure Laser Pro (Experimental): Subjects from the B-Cure Laser Pro group will receive standard care and in addition will self-treat at home daily with the B-Cure device.
  Interventions: Device: B-Cure Laser Pro
- Sham laser (Sham Comparator): Subjects from the Sham laser group will receive standard care and in addition will self-treat at home daily with the sham B-Cure device.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: B-Cure Laser Pro — The B-Cure Laser Pro is a portal, non-invasive low-level laser therapy device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 5J/min
  Arms: B-Cure Laser Pro
Device: Sham laser — The sham laser device is externally identical to the B-Cure Laser Pro and emit the same guiding light, but does not emit the therapeutic near infrared rays
  Arms: Sham laser

SUMMARY:
The global prevalence of diabetes is on the rise and with it increase in prevalence of diabetic foot ulcers (DFU). These recalcitrant wounds are difficult to manage and pose a heavy economic burden. Photobiomodulation (low level laser) is used for acceleration of wound healing. The current study is designed to evaluate the effectiveness of B-cure laser, a home-use low-level laser device, for acceleration of diabetic foot ulcer healing over standard treatment.

DETAILED DESCRIPTION:
Patients with diabetic foot ulcers will receive standard treatment and in addition will be randomly allocated to receive either active or sham laser device to self treat at home. The patient's wound will be evaluated every 2 weeks. Adverse events will be documented. The study hypothesis is that B-Cure laser treatments as an adjunct therapy to standard treatment, applied, at home, by the patient or personal care-giver, can accelerate diabetic foot ulcers healing compared to standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or Female
4. Age:18-95 years old at the time of Informed Consent (Adult, Senior)
5. Type 1 or type 2 Diabetes Mellitus
6. Presence of a diabetic foot ulcer located in the ankle area or below that has persisted a minimum of 3 months prior to the screening visit
7. Ulcer grade classified as ≥2 according to Wagner grading system.
8. Area of ulcer (after debridement) is at least 2 cm2
9. Arterial perfusion: Patients who demonstrate adequate arterial perfusion defined as either: Ankle/brachial index (ABI) above 0.5 or that have documented confirmation of adequate arterial perfusion
10. Patient and/or caregiver must be able and willing to learn and perform the duties of dressing changes
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Exclusion Criteria:

1. Pre-existing conditions - active malignancy,
2. Anemia (Hb<8 gr/dL)
3. Scheduled to undergo vascular surgery, angioplasty, or thrombolysis at the time of enrollment.
4. History of malignancy on study limb or currently receiving or has received radiation or chemotherapy within 3 months of randomization
5. Taking immunosuppressive medication
6. Received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of screening
7. HbA1c > 12% (uncontrolled hyperglycemia)
8. A documented history of alcohol or substance abuse within 6 months of screening
9. Currently enrolled or who have participated, within 30 days of screening, in another investigational device, drug or biological trial that may interfere with study results
10. Pregnant at the time of screening
11. Has any photobiomodulation (low level laser) device at home

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete (100%) wound closure | Up to 3 months
  Complete re-epithelialization without drainage

SECONDARY OUTCOMES:
Time to complete (100%) wound closure | Up to 3 months
  Time to complete re-epithelialization without drainage

CONTACTS AND LOCATIONS:
Overall Officials: Rose Raizman, MSc, MScN, Principal Investigator — Scarborough Health Network
Locations (1):
- Scarborough Health Network ; Centenary Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No